CLINICAL TRIAL: NCT05009823
Title: The Underlying Causes Affecting the Response to Dietary Rehabilitation in Severely Acutely Malnourished Children at the Center Hôspitalier Universitaire Sourô Sanou, Bobo Dioulasso, Burkina Faso
Brief Title: Dietary Rehabilitation in Severely Acutely Malnourished Children
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University Hospital Sourô Sanou of Bobo Dioulasso (Burkina Faso) (Unknown); Centre Muraz (Other)
Responsible Party: Sponsor
Other Study IDs: BC-09443
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Severe Acute Malnutrition; Kwashiorkor; Nutritional Edema; Marasmus
Keywords: Severe acute malnutrition; Nutritional rehabilitation; F75; F100; Ready to use therapeutic food (RUTF); Stabilization phase; Transition phase; Kwashiorkor; Marasmus
MeSH Terms: conditions — Severe Acute Malnutrition; Kwashiorkor; Protein-Energy Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stabilization phase: The dietetic treatment is given by the nurses every 2 hours on the first day; then if tolerance is good, every 3 hours the following days. No family meals during the stabilization phase. But the baby can breastfeed.
  A child will receive an antibiotic as per the national protocol, malaria treatment if diagnosed with malaria, Vitamin A if symptomatic eye damage, Folic acid in case of anemia, antifungal in case of candidiasis.
  Interventions: Dietary Supplement: Standard F75; Dietary Supplement: Alternative F75 With CMV; Dietary Supplement: Alternative F75 Without CMV
- Transition phase: The child is assigned to one the therapeutic regimen depending on the treatment received during the stabilization phase and the results of the appetite test.
  Interventions: Dietary Supplement: F100; Dietary Supplement: Standard F75 + RUTF; Dietary Supplement: Alternative F75 with CMV + RUTF; Dietary Supplement: Alternative F75 without CMV + RUTF

INTERVENTIONS:
Dietary Supplement: Standard F75 — F-75 contains 75 kcal and 0.9 g protein per 100 ml.
  Groups: Stabilization phase
Dietary Supplement: Alternative F75 With CMV — Cereal flour, oil, sugar, powdered milk with complex mineral-vitamin.
  Groups: Stabilization phase
Dietary Supplement: Alternative F75 Without CMV — Cereal flour, oil, sugar, powdered milk without complex mineral-vitamin.
  Groups: Stabilization phase
Dietary Supplement: F100 — 100 kcal and 3 g protein per 100 ml if the test of appetite at the end of the stabilization phase is negative (the child does not accept the Plumpynut)
  Groups: Transition phase
Dietary Supplement: Standard F75 + RUTF — Standard F75 with ready to-use therapeutic food (Plumpynut) if the test of appetite at the end of the stabilization phase is positive
  Groups: Transition phase
Dietary Supplement: Alternative F75 with CMV + RUTF — Alternative F75 + CMV with ready to-use therapeutic food (Plumpynut) if the test of appetite at the end of the stabilization phase is positive and the child received Alternative F75 + CMV during the stabilization phase
  Groups: Transition phase
Dietary Supplement: Alternative F75 without CMV + RUTF — Alternative F75 - CMV with ready to-use therapeutic food (Plumpynut) if the test of appetite at the end of the stabilization phase is positive and the child received Alternative F75 - CMV during the stabilization phase
  Groups: Transition phase

SUMMARY:
Severe acute malnutrition (SAM) is a life threatening condition and is defined by 1) a weight-for-height Z-score more than three standard deviations (SD) below the median based on the 2006 World Health Organization (WHO) growth standards, 2) a mid-upper arm circumference (MUAC) of less than 115 mm or 3) by the presence of nutritional edema. Signs such as edema, mucocutaneous changes, hepatomegaly, lethargy, anorexia, anemia, severe immune deficiency and rapid progression to mortality characterize a state commonly coined as "complicated SAM". Kwashiorkor is one of the forms of complicated SAM commonly distinguished by the unmistakable presence of bipedal edema. SAM results in high mortality rates of up to half a million child deaths annually. Undernourished children are at higher risk of mortality ranging from three-times more risk among children with moderate malnutrition to 10-times in SAM children compared to well-nourished children. Children with complicated SAM require inpatient treatment in specialized centers.

The "Rehabilitation and Nutritional Education Center" (CREN) is a specialized center in Burkina Faso receiving on average 10 SAM children per day. Recovery rate is lower than international standards; and adverse events and mortality remain strikingly high.

The main objective of this study is to assess the underlying risk factors affecting the effectiveness of the nutritional therapeutic treatment protocol for complicated SAM children under 5 years of age who have been referred to the CREN, at the Centre Hôspitalier Universitaire Souro, Bobo Dioulasso, Burkina Faso.

The specific objective of this study is to better understand underlying risk factors associated with a lower recovery rate and high mortality in complicated SAM children referred to CREN for inpatient care. Risk factors associated with poor response to a standard dietary treatment at any phase will be assessed retrospectively.

DETAILED DESCRIPTION:
Severe acute malnutrition (SAM), defined as severe wasting [weight-to-height Z-score < -3 standard deviations (SD), based on the WHO Child Growth Standards] and / or the presence of nutritional edema, and / or mid-upper arm circumference (MUAC) <115 mm, is a condition that requires urgent attention and appropriate management to reduce mortality and promote recovery among children. Management of SAM children without complications is provided at the community level. Hospitalization in specialized care centers is necessary for SAM children with complications. SAM children with comorbidities have a greater risk of mortality and treatment failure. The knowledge of the specific adequate nutritional needs of SAM is limited.

For the treatment of SAM in hospital, the WHO recommends the use of therapeutic milk low in protein 'F75' in the stabilization phase; and more protein-rich F100 or F75 combined with ready-to-use therapeutic foods (RUTF) in the transition phase. The WHO also recommends using as an alternative formula made of cereal flour, skimmed milk powder, oil, sugar, and a therapeutic vitamin and mineral complex (CMV), in case of shortage of the standard therapeutic milk F75 / F100 or in case of signs of intolerance (vomiting, diarrhea).

The Refeeding Center - Centre de Récupération et d'Education Nutritionnelle (CREN) of the Sourô Sanou University Hospital Center (CHUSS) in Burkina Faso specializes in the care of SAM children with complications. In 2018, out of 500 children aged 6-59 months admitted for SAM with complications, the CHUSS CREN registered 86.8% full recovery, 8.2% dropout and 5% death. Although the recovery rate is higher than international standards (greater than 75%), the mortality rate remains higher than the recommended 3% by international standards; in addition to the challenges that are faced locally in maintaining high standards of care. At the CREN, the investigators and the nurses observed that some SAM children with complications can have severe diarrhea and vomiting after taking F75 (first phase of the nutritional treatment). It was also observed that other SAM children with edema, whose edema resolved in the first phase of treatment under F75, redeveloped edema when they received RUTF (Plumpy Nut®) in the transition phase according to the WHO 2013 protocol.

This research project, which will be subdivided into a retrospective study and two prospective clinical trials aims to assess the risk factors affecting the response to dietary treatment in this center (the CREN, Burkina Faso) and to compare alternatives for treatment during the nutritional rehabilitation.

The retrospective study assesses the factors of failure of dietary treatment in the three phases of nutritional rehabilitation to better understand underlying risk factors associated with a lower recovery rate and high mortality in complicated SAM children referred to CREN for inpatient care. Risk factors associated with poor response to a standard dietary treatment at any phase will be assessed retrospectively and include:

1. Errors in the treatment (feeding) dosage that can be due to errors in anthropometric measurement and/or in reading the feeding regimen table by the CREN team;
2. Low adherence of children to the therapeutic dietary regimen
3. Comorbidities associated with malnutrition that can have an effect on the dietary treatment effectiveness
4. Types of dietary regimen selected during the first phase of treatment [F75 vs. alternative F75 (cereal flour, oil, sugar, powdered milk) with OR without CMV)] and during the transition phase [F75 + RUTF ( Plumpy-Nut®), F100, alternative F75 (with and without CMV) + RUTF (Plumpy Nut®)].

The study will use data collected during admission and follow-up of SAM children with complications admitted at the CREN of the CHUSS from January 2014 to December 2018.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute malnutrition defined as Weight-for-Height Z-score (WHZ) <- 3 SD AND / OR MUAC <115 mm AND / OR with edema
* With complications
* Who were admitted and treated in the refeeding center (CREN) of the CHUSS from January 2014 TO December 2018
* Aged between 0 and 59 Months

Exclusion Criteria:

* Older than 59 Months
* Moderate Acute Malnutrition (MAM)

Ages: 0 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible participants are children 0-59 Months of age who were hospitalized in the pediatric department for SAM with or without edema, and children hospitalized in other departments from CHUSS and received at CREN for treatment of SAM.
Sampling Method: Non-Probability Sample
Enrollment: 1959 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of days during the first phase of treatment | Three to Seven days
  Average number of days spent in the stabilization phase in Days
Number of days during the transition phase of treatment | Three to Five days
  Average number of days spent in the transition phase in Days
Daily weight gain during the first phase of treatment | Three to Seven days
  Average daily weight gain in the stabilization phase in Grams
Daily weight gain during the transition phase | Three to Five days
  Average daily weight gain in the transition phase in Grams
Edema redevelopment during the transition phase | Three to Five days
  Edema redevelopment during the transition phase after starting to resolve during the stabilizing phase.

SECONDARY OUTCOMES:
Anorexia | Through study completion, an average of 15 days
  Serious severe event that occurs at anytime during the treatment
Mortality | Through study completion, an average of 15 days
  Serious severe event that occurs at anytime during the treatment
Diarrhea | Through study completion, an average of 15 days
  Serious severe event that occurs at anytime during the treatment
Vomiting | Through study completion, an average of 15 days
  Serious severe event that occurs at anytime during the treatment
Adherence to the dietary treatment | Through study completion, an average of 15 days
  Daily intake of the administered dietary treatment

OTHER OUTCOMES:
HIV/AIDS | Through study completion, an average of 15 days
  Detection of HIV/AIDS using polymerase chain reaction (PCR) in infants and children younger than 18 months or retroviral serology test in older children
Hepatitis | Through study completion, an average of 15 days
  Test of hepatitis
Tuberculosis | Through study completion, an average of 15 days
  Test of tuberculosis
Tumoral pathologies (benign or malignant) | Through study completion, an average of 15 days
  Clinical diagnosis
Malformative pathologies | Through study completion, an average of 15 days
  Clinical diagnosis
Diabetes | Through study completion, an average of 15 days
  Clinical diagnosis
Renal failure. | Through study completion, an average of 15 days
  Clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent; Jerome Some, Md. PhD, Principal Investigator — Institut de Recherche en Sciences de la Sante, Burkina Faso; Bintou Sanogo, MSc. Md., Principal Investigator — Centre Hospitalier Universitaire Souro, Bobo Dioulasso, Burkina Faso.
Locations (1):
- Centre Hospitalier Universitaire Souro, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: No
All the data that can affect the main or the secondary outcomes will be used in the analyses and shared as necessary.

REFERENCES:
- [Background] Baraki AG, Akalu TY, Wolde HF, Takele WW, Mamo WN, Derseh B, Desyibelew HD, Dadi AF. Time to recovery from severe acute malnutrition and its predictors: a multicentre retrospective follow-up study in Amhara region, north-west Ethiopia. BMJ Open. 2020 Feb 13;10(2):e034583. doi: 10.1136/bmjopen-2019-034583. PMID 32060161
- [Background] Bartz S, Mody A, Hornik C, Bain J, Muehlbauer M, Kiyimba T, Kiboneka E, Stevens R, Bartlett J, St Peter JV, Newgard CB, Freemark M. Severe acute malnutrition in childhood: hormonal and metabolic status at presentation, response to treatment, and predictors of mortality. J Clin Endocrinol Metab. 2014 Jun;99(6):2128-37. doi: 10.1210/jc.2013-4018. Epub 2014 Feb 27. PMID 24606092
- [Background] Deen JL, Funk M, Guevara VC, Saloojee H, Doe JY, Palmer A, Weber MW. Implementation of WHO guidelines on management of severe malnutrition in hospitals in Africa. Bull World Health Organ. 2003;81(4):237-43. Epub 2003 May 16. PMID 12764489
- [Background] Munthali T, Jacobs C, Sitali L, Dambe R, Michelo C. Mortality and morbidity patterns in under-five children with severe acute malnutrition (SAM) in Zambia: a five-year retrospective review of hospital-based records (2009-2013). Arch Public Health. 2015 May 1;73(1):23. doi: 10.1186/s13690-015-0072-1. eCollection 2015. PMID 25937927
- See also: World Health Organization (2013) WHO guideline: updates on the management of severe acute malnutrition in infants and children. — https://www.who.int/publications/i/item/9789241506328
- See also: Enquête Nutritionnelle Nationale SMART 2016 au Burkina Faso. 2016 ; 47p. — https://www.unicef.fr/article/malnutrition-la-situation-au-burkina-faso
- See also: 10. Ministère de la Sante au Burkina Faso. Protocol National : Prise en charge intégrée de la malnutrition aigüe (PCIMA). 2014 — https://www.humanitarianresponse.info/sites/www.humanitarianresponse.info/files/documents/files/protocole_pcima_bf_janv_2015.pdf